CLINICAL TRIAL: NCT04636710
Title: Refining Local-Regional Therapy for Inflammatory Breast Cancer (IBC)
Brief Title: Refining Local-Regional Therapy for IBC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Faina Nakhlis, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-151
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Inflammatory Breast Cancer; Sentinel Lymph Node
Keywords: Breast Cancer; Inflammatory Breast Cancer; Sentinel Lymph Node
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sentinal Node Identification (Experimental): Within standard of care treatment for inflammatory breast cancer, participants will undergo a series of Lymphoscintigraphies: an imaging procedure to determine where their lymphatic system drains from their breast.
  * Prior to neoadjuvant chemotherapy
  * Day before surgery
  These two imaging studies will be compared and the information used during participant's surgery to perform the sentinel node biopsy procedure.
  During surgery participants will have a blue dye injected to affected breast to map drainage and identify sentinal nodes. The sentinal nodes will be removed first, followed by standard of care procedure to remove all axillary lymph nodes.
  After surgery, a small amount of tissue from the tumor removed during surgery will be evaluated.
  Participants will complete a Lymphedema Questionnaire after each Lymphoscintigraphy then every 6 months for 2 years post surgery.
  Interventions: Procedure: Lymphoscintigraphy

INTERVENTIONS:
Procedure: Lymphoscintigraphy — An imaging procedure using an injected radioactive substance or dye to identify lymph drainage A doctor reviews the images to identify the sentinel lymph nodes based on where the dye goes to first.
  Other Names: Sentinel lymph node mapping

SUMMARY:
This Feasibility study is trying to determine:

* If Lymphoscintigraphy (imaging of the lymphatic drainage patterns) is effective in demonstrating the drainage to the sentinel lymph nodes in patients with inflammatory breast cancer.
* The likelihood of identifying the sentinel lymph nodes in the operating room, using both blue dye and the radioactive substance used for lymphoscintigraphy.
* The incidence of lymphedema (arm swelling which occurs after lymph node surgery) in women with inflammatory breast cancer
* Outcomes for women with inflammatory breast cancer, whether or not the sentinel lymph nodes can be identified.

DETAILED DESCRIPTION:
This research study is a Feasibility Study, which means the investigators are collecting information from a relatively small group of patients to determine if the sentinel lymph node procedure identifies the first nodes that drain the breast in patients with inflammatory breast cancer.

The sentinel node procedure is a standard method to evaluate whether breast cancer has spread to the axillary lymph nodes (lymph nodes under the arm) or remains in the lymph nodes under the arm after chemotherapy in non-inflammatory breast cancer. "Standard" means that sentinel lymph node biopsy is accepted by the majority of the medical community as a suitable method to determine if breast cancer has spread to the lymph nodes or remains in the lymph nodes after chemotherapy. In women with non-inflammatory breast cancer, these lymph nodes are tested first and if they are free of cancer additional lymph nodes are not removed. By safely limiting the amount of lymph node surgery to only the sentinel lymph nodes, the likelihood of developing lymphedema (arm swelling after lymph node surgery) has declined among women with non-inflammatory breast cancer.

Currently, sentinel lymph node biopsy is not performed in inflammatory breast cancer as there are little data supporting that it works or is accurate. For inflammatory breast cancer, performing lymphoscintigraphy (imaging study to show the drainage from the breast to the lymph nodes) and sentinel lymph node biopsy is investigational. "Investigational" means that this is being studied. If in this study it is determined that sentinel lymph nodes can be accurately identified and tested in patients with inflammatory breast cancer, this could lead to future studies testing whether complete lymph node dissection can be avoided in women with inflammatory breast cancer whose sentinel nodes are free of cancer. Thus, potentially also reducing the likelihood of lymphedema in patients who receive treatment for inflammatory breast cancer.

The research study procedures include screening for eligibility, imaging evaluation, lymphoscintigraphy, sentinel lymph node evaluation, a mandatory research biopsy, research blood draws and questionnaires.

It is expected that about 50 people will take part in this research study at participating sites around the United States

Johns Hopkins University on behalf of the Translational Breast Cancer Research Consortium (TBCRC) is supporting this research study by providing funding for the research study. The TBCRC is a group of academic medical centers across the United States that work together to conduct breast cancer research.

ELIGIBILITY:
Inclusion Criteria:

* Stage III IBC (cT4d cN0-2). Inflammatory breast cancer is defined as the following constellation of symptoms (all of the following must be met):

  * Rapid onset symptoms (6 months or less from time of diagnosis)
  * Breast erythema, edema and/or peau d'orange and/or warm breast with or without an underlying palpable mass
  * Erythema occupying at least one-third of the breast
  * Pathologic confirmation (biopsy-proven) invasive breast carcinoma
* Women age ≥18 years
* ECOG performance status ≤2
* Ability to understand and willingness to sign informed consent document and comply with study procedures, including baseline research biopsy. If the research biopsy is not felt to be reasonably safe or feasible, a waiver must be obtained from the Principal Investigator. A formal exception would not be required in this case.

Exclusion Criteria:

* Participants who initiated pre-operative/neoadjuvant therapy prior to registration are ineligible.
* Participants with Stage IV (metastatic) breast cancer are excluded. The absence of any evidence of distant disease on staging studies needs to be confirmed at the time of diagnosis (within 42 days from initial presentation) using the staging studies that are standard for the participating institution.
* Participants with positive contralateral axillary nodes identified on standard imaging studies (MMG, MRI, US) are excluded. In participants with clinically suspicious axillary nodes, US guided biopsy will be performed prior to registration. If the contralateral axillary biopsy is positive, patients will not be eligible. If standard imaging does not identify contralateral disease yet drainage to the contralateral axillary basin is identified on pre-NAC lymphoscintigraphy, contralateral axillary US (if not already performed) will be obtained and any suspicious contralateral axillary nodes will undergo US guided biopsy. If the contralateral axillary biopsy is positive, patients will not continue on study for the evaluation of the primary endpoint, but their data will be used for the descriptive analyses of lymphatic drainage patterns in IBC. Contralateral invasive breast cancer without axillary involvement or in-situ carcinoma in either breast is allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Sentinel Lymph Node (SLN) identification rate | Up to 6 months
  The identification rate will be calculated as a ratio of the number of patients in whom SLN(s) were successfully identified over the total number of patients in whom SLN mapping was attempted.

SECONDARY OUTCOMES:
Prevalence of lymphedema | Every 6 months post surgery up to 2 years
  Assess the prevalence of lymphedema following comprehensive local therapy (surgery + regional RT) using the patient-reported Lymphedema Symptom Intensity and Distress Survey - Arm (LSIDS-A) (Appendix A).
Local-regional recurrence free survival rate (LRRFS) | Within 2 years from surgery
  Duration of time from surgery until invasive ipsilateral local-regional recurrence or death from any cause; in the absence of an event, LRRFS will be censored at the date last know alive and free from local regional recurrence (LRR).
Distant recurrence-free survival rate (DRFS) | Within 2 years from surgery
  Duration of time from surgery until distant recurrence or death from any cause; in the absence of an event, DRFS will be censored at the date last know alive and free from distant recurrence
Disease-free survival (DFS) | Within 2 yhears from surgery
  Duration of time from surgery until invasive ipsilateral local regional recurrence, invasive contralateral breast cancer, distant recurrence, or death from any cause; in the absence of an event, DFS will be censored at the date last know alive and free from all events.

CONTACTS AND LOCATIONS:
Overall Officials: Faina Nahklis, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu